CLINICAL TRIAL: NCT06540729
Title: Disitamab Vedotin (RC48) in Combination With AK104 (PD-1/CTLA-4 Bispecific) and Bevacizumab for the Treatment of Recurrent and Persistent Clear Cell Ovarian Cancer
Brief Title: RC48 in Combination With AK104 and Bevacizumab in OCCC
Acronym: DAB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-532-01
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-08

CONDITIONS: Ovary Cancer
Keywords: Disitamab vedotin; AK104; bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — disitamab vedotin; Bevacizumab

STUDY DESIGN:
Intervention Model Description: we are initiating this clinical study aimed at evaluating the efficacy and safety of vedolizumab (HER2-targeted ADC) in combination with AK104 (anti-PD-1 and CTLA4) and bevacizumab (anti-angiogenesis) in recurrent and persistent OCCC patients (vedolizumab 2.5 mg/kg + AK104 10 mg/kg + bevacizumab 15 mg/kg, every 3 weeks), with the aim of providing new treatment options for these refractory gynecologic malignancies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Disitamab vedotin (RC48) in combination with AK104 (PD-1/CTLA-4 bispecific) and bevacizumab for the treatment of recurrent and persistent clear cell ovarian cancer
  Interventions: Drug: Disitamab vedotin in combination with AK104 and bevacizumab for the treatment of recurrent and persistent clear cell ovarian cancer

INTERVENTIONS:
Drug: Disitamab vedotin in combination with AK104 and bevacizumab for the treatment of recurrent and persistent clear cell ovarian cancer — Disitamab vedotin (RC48) in combination with AK104 (PD-1/CTLA-4 bispecific) and bevacizumab for the treatment of recurrent and persistent clear cell ovarian cancer

SUMMARY:
Disitamab vedotin (RC48) in combination with AK104 (PD-1/CTLA-4 bispecific) and bevacizumab for the treatment of recurrent and persistent clear cell ovarian cancer: a single-arm, phase II, multicenter study (DAB OCC study)

DETAILED DESCRIPTION:
Ovarian clear cell carcinoma (OCCC) ranks as the second most common epithelial ovarian malignancy in Asian women, characterized by extremely poor prognosis, with a median overall survival (OS) of 25.3 months. OCCC demonstrates a dismal response rate to conventional chemotherapy, and once in a state of persistence or recurrence, treatments become severely limited, with a mere 5-year survival rate of 13.2%, with over two-thirds of patients succumbing within 1 year. Thus, there is an urgent need to explore new therapeutic approaches for recurrent and persistent OCCC patients. Evidence suggests that anti-angiogenesis therapy is effective against OCCC, which tends to exhibit a "hot tumor" phenotype. Hence, the combination of anti-angiogenesis therapy with immunotherapy holds promise for recurrent and persistent OCCC. Additionally, overexpression of human epidermal growth factor receptor 2 (HER2) plays a pivotal role in OCCC resistance formation. Antibody drug conjugates (ADCs) targeting HER2 have shown increasing efficacy in ovarian cancer treatment, with significant immunomodulatory effects enhancing the efficacy of immunotherapy. Based on this evidence, the investigators hypothesize that the combination of anti-angiogenesis therapy, immunotherapy, and HER2-targeted ADCs may improve the prognosis of OCCC patients. Therefore, the investigators are initiating this clinical study aimed at evaluating the efficacy and safety of vedolizumab (HER2-targeted ADC) in combination with AK104 (anti-PD-1 and CTLA4) and bevacizumab (anti-angiogenesis) in recurrent and persistent OCCC patients (vedolizumab 2.5 mg/kg + AK104 10 mg/kg + bevacizumab 15 mg/kg, every 3 weeks), with the aim of providing new treatment options for these refractory gynecologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis confirms ovarian clear cell carcinoma. In cases of mixed carcinoma, a prerequisite is that clear cell carcinoma constitutes at least 70% of the tumor mass. Moreover, adherence to RECIST 1.1 criteria mandates the presence of at least one evaluable lesion.
* HER2 IHC ≥1+.
* Treatment-naïve individuals encompass those experiencing tumor progression during postoperative chemotherapy and those who, following platinum-containing neoadjuvant chemotherapy, have not undergone surgical intervention yet and subsequently manifested progression during or after platinum-containing chemotherapy, provided that they have received a maximum of 2 prior lines of chemotherapy.
* Recurrent patients, whether platinum-sensitive or platinum-resistant, include those lacking a platinum-free interval of ≥6 months and who, post-recurrence, have undergone re-administration of platinum-containing chemotherapy but have demonstrated an inability to tolerate toxic reactions, with a maximum of 2 lines of chemotherapy post-recurrence.
* Previous utilization of bevacizumab is permissible.
* Adequate bone marrow reserve function necessitates pre-operative blood routine parameters meeting specific criteria: white blood cell count ≥3.0×10^9/L, neutrophil count ≥1.5×10^9/L, platelet count ≥100×10^9/L, and hemoglobin ≥80 g/L.
* atisfactory organ function entails biochemical test results within defined limits: AST ≤2.5× upper limit of normal (ULN), ALT ≤2.5× ULN, serum total bilirubin ≤1.5× ULN, and creatinine ≤1.5× ULN.
* ECOG performance status score ranging from 0 to 1.
* Patient participation is contingent upon voluntary execution of an informed consent form.

Exclusion Criteria:

* Patients with a history of immunotherapy, including treatments targeting PD-1, PD-L1, CAR-T, and CTLA-4.
* Patients diagnosed with other malignancies within the past five years, excluding skin cancer and thyroid cancer.
* Patients with an expected survival of ≤12 weeks.
* Patients with a known allergy to taxane-based medications.
* Patients who, based on clinical assessment, have contraindications for receiving immunotherapy and/or bevacizumab, such as uncontrolled infections, gastrointestinal fistula, autoimmune diseases, active hepatitis, or active bleeding.

Patients currently undergoing treatment with investigational anti-cancer drugs in other clinical trials.

* Patients with any unstable condition or situation that may compromise their safety or adherence to the study protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  Objective response rate of advanced or recurrent ovarian clear cell carcinoma

SECONDARY OUTCOMES:
Time to progress | 2 years
  Time to progress of advanced or recurrent ovarian clear cell carcinoma
Adverse event | 2 years
  Adverse event rate of treatment with RC48 in combination with AK104 and bevacizumab
The time to the first subsequent therapy | 2 years
  The time to the first subsequent therapy for enrolled patients
Time to response | 2 years
  Time to response for enrolled patients
Duration of response | 2 years
  Duration of response of advanced or recurrent ovarian clear cell carcinoma
Disease control rate | 2 years
  Disease control rate of patients with recurrent or advanced ovarian clear cell carcinoma receiving intervention
Progression free survival | 2 years
  Progression free survival of enrolled patients with recurrent or advanced ovarian clear cell
Overall survival | 2 years
  Overall survival of enrolled patients with recurrent or advanced ovarian clear cell
Eastern Cooperative oncology group performance status score | 2 years
  ECOG score of enrolled patients

OTHER OUTCOMES:
Biomarker | 2 years
  Explore biomarkers for predicting the response of OCCC to combination therapy, including but not limited to PD-L1, TMB, MMRd, MSI-H, HRR related genes, and lymphocyte infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Don't share IPD